CLINICAL TRIAL: NCT00545766
Title: A Phase II Trial of Vinflunine as Salvage Chemotherapy in Hormone Refractory Prostate Cancer (HRPC)
Brief Title: Vinflunine in Hormone Refractory Prostate Cancer (HRPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 35
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Hormone Refractory; Vinflunine; Salvage Chemotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interventional (Experimental)
  Interventions: Drug: Vinflunine

INTERVENTIONS:
Drug: Vinflunine — Vinflunine 320 mg/m2 will be administered as a 20 minute IV infusion q3w. Patients will be evaluated for toxicity after each cycle of therapy. Response to vinflunine will be assessed every 6 weeks (every 2 cycles) of treatment. A maximum of 6 cycles of therapy are planned.
  Other Names: Javlor

SUMMARY:
Currently, there are no established 2nd-line or salvage chemotherapy regimens for patients with HRPC, many of whom retain an excellent performance status. The antitumor characteristics and toxicity profile of vinflunine make it an ideal agent to be investigated in this setting. In this Phase II trial, we plan to evaluate the efficacy, toxicity, and feasibility of administering IV vinflunine at a dose of 320 mg/m2 q3w as salvage chemotherapy in patients with HRPC. The patients will be evaluated for response, survival, and toxicity. If significant antitumor activity is demonstrated, further evaluation of this agent either alone or combination regimens and at earlier stages of disease will be indicated.

DETAILED DESCRIPTION:
This is a non-randomized (single-arm), open-label, multi-center, single-agent, Phase II study of vinflunine as second- or third-line treatment of subjects with HRPC. The primary objective of the study is to evaluate the efficacy of vinflunine in the salvage treatment, as measured by Protein-Specific Antigen (PSA) Response Rate endpoint.

The primary objective of this study is as follows:

To evaluate the efficacy (as measured by the PSA response rate) of IV vinflunine administered q3w in HRPC patients who have progressed after one or two previous chemotherapy regimens.

Secondary Objectives

The secondary objectives of this study are as follows:

* To evaluate the efficacy of IV vinflunine administered q3w in HRPC patients who have previously received chemotherapy (one or two regimens), as measured by:

  * Time to PSA progression
  * Overall survival
  * Palliative response in patients with an Analgesic Score (AS) ≥10 and stable baseline pain
  * Health-Related Quality of Life
* To assess the efficacy (as measured by the PSA response rate) of IV vinflunine in HRPC patients based on their response to prior chemotherapy
* Chemotherapy responsive - previous response to most recent chemotherapy regimen lasting >2 months after completion.
* Chemotherapy refractory - failure to respond to, or progression during or within three months of completing last chemotherapy.
* To assess the response rate to IV vinflunine in the subset of patients with measurable disease, as measured by traditional Response Evaluation Criteria in Solid Tumors (RECIST) criteria (Therasse et al. 2000).
* To evaluate the safety of IV vinflunine administered every three weeks in HRPC patients who have previously received chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Men age 18 years of age or older who have HRPC are eligible for this study based on the following inclusion criteria:

1. Histologically confirmed adenocarcinoma of the prostate.
2. Progressive hormone refractory locally advanced or metastatic disease.

   * (Definition of HRPC): Clinical or serological evidence of disease progression despite adequate anti-androgen therapy, documented by castrate levels of serum testosterone (<50 ng/mL).
   * Patients on medical castration therapy should continue on treatment to maintain castrate levels of serum testosterone. Patients receiving anti-androgen or estrogen therapy should either be maintained on it, or have documented progression 4 weeks after withdrawal of all agents (except nilutamide and bicalutamide), which requires 6 weeks.
3. Disease Progression, documented by any of the following:

   * PSA Progression, documented by an elevated PSA level (>5 ng/mL), which has risen serially from the baseline PSA value (PSA value #1) on two occasions, each at least 1 week apart (these will be considered PSA values #2 and #3). (Note: if the level of PSA value #3 is less than the level of PSA value #2, a subsequent PSA value must be obtained (PSA value #4) at least 1 week after PSA value #3 was measured. In order for this event to be considered a PSA progression, the level of this final PSA value (PSA value #4) must be greater than the PSA level that was observed for PSA value #2.
   * Progressive metastatic prostate carcinoma, documented by computed tomography (CT), magnetic resonance imaging (MRI), or radiograph of non osseous lesions (see Section 7.2).
   * Bone Scan Progression, documented by the appearance of at least one or more new lesions that are not believed to be secondary to tumor flare phenomenon.
4. Patients with bone only disease must have a PSA level >=5 ng/mL; patients with stable lesions must have evidence of PSA progression. Patients must have radiographically or clinically demonstrable metastatic disease.
5. Receipt of either 1 or 2 previous chemotherapy regimens; one of these regimens must have included docetaxel.
6. ECOG performance status of 0-2.
7. Adequate bone marrow function, defined by: white blood cells >=3,500/uL, hemoglobin >=8 g/dL, platelet count >=100,000/uL.
8. Adequate renal function, defined by: serum creatinine <1.8 mg/dL, or calculated or measured creatinine clearance (GFR) of >=60 cc/min. Patients with a creatinine clearance of >30 mL/min but <60 mL/min may also be enrolled, but will require an initial adjusted dose (see Section 5.1)
9. Adequate hepatic function, defined by: total bilirubin <1.5 x the upper limit of normal, AST <2 x the upper limit of normal.
10. Patients must be able to comprehend the nature of the study and provide written informed consent.
11. Partners of women of childbearing potential must use effective contraception while on treatment and for at least 3 months thereafter. Women of childbearing potential include females who have experienced menarche and have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not post-menopausal (i.e., amenorrhea >12 months).
12. Patients on bisphosphonate therapy (at the discretion of the investigator).

Exclusion Criteria:

1. History of other prior malignancy in the past 5 years (excluding resected basal cell or squamous cell skin cancer).
2. History of second- or third-degree heart block, uncontrolled angina, uncontrolled hypertension, or recent myocardial infarction or congestive heart failure (New York Heart Association Class III-IV) within the past 6 months (see Appendix F)
3. Cerebral vascular accident within the past 6 months.
4. Peripheral neuropathy > grade 2 per Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
5. Patients with rising PSA but no demonstrable metastases.
6. Previous radiotherapy, outside of standard portals, utilized for prostate cancer (if total amount of radiotherapy encompasses >25% of bone marrow containing osseous regions).
7. Prior therapy with Strontium 90, Samarium 150, or other injectable therapeutic radioisotopes.
8. History of prior allergic reaction to any vinca alkaloid.
9. Use of chemotherapy or investigational drugs within 4 weeks prior to the first dose of study drug.
10. Treatment with ketoconazole, itraconazole, ritonavir, amprenavir, or indinavir within 4 weeks prior to the first dose of study drug.
11. Previous treatment with an anthracycline.
12. Patients who are unable to receive chemotherapy on a basis of once every three weeks as a result of physical, environmental, or co existent medical problems.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-05; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (12):
- United States (12):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Oncology Hematology Care, Cincinnati, Ohio
  - Consultants in Medical Oncology and Hematology, Drexel Hill, Pennsylvania
  - Associates in Hematology Oncology, Chattanooga, Tennessee
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Peninsula Cancer Institute, Newport News, Virginia

REFERENCES:
- [Result] Hainsworth JD, Meluch AA, Lane CM, Spigel DR, Burris HA 3rd, Gandhi JG, Crane EJ, Stipanov MA, Greco FA. Single agent vinflunine in the salvage treatment of patients with castration-resistant prostate cancer: a phase II trial of the Sarah Cannon research consortium. Cancer Invest. 2010 Mar;28(3):275-9. doi: 10.3109/07357900902918460. PMID 20158340

RESULTS

PARTICIPANT FLOW:
Groups:
- Vinflunine: Vinflunine : Vinflunine 320 mg/m2 will be administered as a 20 minute IV infusion q3w. Patients will be evaluated for toxicity after each cycle of therapy. Response to vinflunine will be assessed every 6 weeks (every 2 cycles) of treatment. A maximum of 6 cycles of therapy are planned.
Period: Overall Study
Arm/Group | Vinflunine
Started | 41
Completed | 36
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Vinflunine
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Protein-specific Antigen (PSA) Response Rate
Description: Defined as the percentage of patients with an objective decrease in PSA and/or experience an objective benefit from treatment.
Time Frame: 18 months
Population: Five patients did not receive two full cycles of vinflunine and were not included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vinflunine
Number analyzed (Participants) | 36
percentage of patients | 3 [-2.57 to 8.57]

2. Secondary Outcome: Time to PSA Progression
Description: Time to PSA Progression is defined as the time from the first dose administration to the date when criteria for PSA progression (for Progressive Disease) are initially met.
Time Frame: 18 months
Population: 38 patients with serial PSA evaluations were included in the analysis. 3 patients only had baseline evaluations and were not included in analysis.
Measure: Mean (Full Range); unit: weeks
Arm/Group | Vinflunine
Number analyzed (Participants) | 38
weeks | 12.2 [2.7 to 57.1]

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time from the first day of treatment until the day tumor progression was documented. Response categories were assigned after completion of two weeks of vinflunine therapy using Response Evaluation Criteria in Solid Tumors (RECIST). Progressive disease is defined as an increase in >=25% of of serum PSA above baseline value documented by at least two successive values separated by at least one week.
Time Frame: 18 months
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Vinflunine
Number analyzed (Participants) | 36
months | 2.1 [1.4 to 2.9]

4. Secondary Outcome: Number of Participants Experiencing Overall Survival (OS)
Description: OS is defined as the time from the first treatment until date of death due to any cause. In the absence of confirmation of death or lack of data beyond follow-up period, the survival time was censored to last date the participant was known to be alive. Number of participants experiencing overall survival is reported here.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vinflunine
Number analyzed (Participants) | 41
Participants | 15

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Vinflunine
All-Cause Mortality (participants affected / at risk) | 26/41
Serious Adverse Events (participants affected / at risk) | 11/41
Other Adverse Events (participants affected / at risk) | 33/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vinflunine (N=41)
Pain - abdomen (General disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Infection - Pneumonia (Infections and infestations) | 1 (1)
Cardiac arrhythmia (Cardiac disorders) | 1 (1) — Arrhythmia not otherwise specified
Cardiac ischemia (Cardiac disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 3 (4)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Pain - back (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vinflunine (N=41)
Abdominal pain (Gastrointestinal disorders) | 9 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (11)
ANC (Blood and lymphatic system disorders) | 30 (50)
Anorexia (Gastrointestinal disorders) | 14 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (20)
Constipation (Gastrointestinal disorders) | 22 (36)
Dehydration (Gastrointestinal disorders) | 3 (6)
Depression (Nervous system disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (14)
Edema (Vascular disorders) | 6 (12)
Fatigue (General disorders) | 33 (72)
Febrile Neutropenia (Infections and infestations) | 4 (5)
Headache (Nervous system disorders) | 5 (9)
HGB (Blood and lymphatic system disorders) | 31 (76)
Hot flashes (Endocrine disorders) | 4 (5)
Infection without Neutropenia (Infections and infestations) | 4 (5)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 7 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (11)
Nausea (Gastrointestinal disorders) | 17 (27)
Pain (General disorders) | 2 (3)
Pain (back) (Musculoskeletal and connective tissue disorders) | 3 (3)
PLT (Blood and lymphatic system disorders) | 13 (21)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Sensory Neuropathy (Nervous system disorders) | 7 (15)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 9 (11)
WBC (Blood and lymphatic system disorders) | 32 (59)
Weakness (General disorders) | 9 (13)
Weight Loss (General disorders) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.